CLINICAL TRIAL: NCT02819778
Title: Interventional Study Assessing Evaluation of the Interest of Serum S100B Protein Determination in the Management of Pediatric Mild Traumatic Brain Injury
Brief Title: Study Assessing Evaluation of the Interest of Serum S100B Protein Determination in the Management of Pediatric Mild Traumatic Brain Injury
Acronym: PROS100B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0269; 2016-A00195-46 (Other: 2016-A00195-46)
Record Dates: First submitted 2016-06-24; First posted 2016-06-30 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2022-05

CONDITIONS: Craniocerebral Trauma; Pediatrics
Keywords: Diagnosis; Craniocerebral Trauma; Pediatrics; S100B; mild traumatic brain injury
MeSH Terms: conditions — Craniocerebral Trauma; Disease; Brain Concussion

ARMS (2):
- Control group (Other): The study protocol corresponds to a diagnostic prospective, controlled, multicenter study using a randomized stepped wedge cluster design, in which pediatric patients (aged ≤ 16 years) presenting to the pediatric emergency room for mTBI with a GCS score of 15 will benefit from usual care ("conventional management" arm) in the control group, and from S100B management in the interventional group
  Interventions: Procedure: usual care
- interventional group (Other): The study protocol corresponds to a diagnostic prospective, controlled, multicenter study using a randomized stepped wedge cluster design, in which pediatric patients (aged ≤ 16 years) presenting to the pediatric emergency room for mTBI with a GCS score of 15 will benefit from usual care ("conventional management" arm) in the control group, and from S100B management in the interventional group
  Interventions: Procedure: S100B

INTERVENTIONS:
Procedure: usual care
  Arms: Control group
Procedure: S100B
  Arms: interventional group

SUMMARY:
Mild traumatic brain injury (mTBI) is a very common reason for presentation to pediatric emergency departments. So as not to overlook the risk of complications, which occur at a rate of 0-7%, measures such as cranial computed tomography (CCT-scan) and/or short inpatient observation are prescribed. Ultimately, the majority of these measures could be avoided and a large Australian cohort shows that the risk of brain tumors is 2.44 times higher for children who had a CCT-scan (3.24 for age 1-4 years). Assay of a sensitive biomarker in blood, such as the S100B protein, has the potential to reduce the number of these unnecessary measures.

DETAILED DESCRIPTION:
Based on initial results from a previous prospective study, a multicenter interventional study will be necessary to validate the routine use of this biomarker .The ultimate goal is to include serum S100B assay in the current recommendations for m traumatic brain injury (mTBI) management based on the study of Kupperman et al. (2009), as mTBI accounts for 5-8% of pediatric emergency admissions in France (60-100 per 100,000 children). The study of Kuppermann et al. strongly dictated the recommendations for mTBI management by the French Society of Emergency Medicine (SFMU) . Then, from these 2 publications, the French Society of Pediatrics (SFP) redacted their recommendations after adjustment method recommendations for clinical practice, used by the French High Authority of Health (HAS) .

The use of serum S100B assay as part of the management of pediatric mTBI should make it possible to reduce the number of additional examinations, in particular a 30% reduction in the number of CCT-scans, with a resultant reduction in radiation exposure, known to be a risk factor for cancer. The study protocol corresponds to a diagnostic prospective, controlled, multicenter study using a randomized stepped wedge cluster design, in which pediatric patients (aged ≤ 16 years) presenting to the pediatric emergency room for mTBI with a GCS score of 15 will benefit from usual care ("conventional management" arm) in the control group, and from S100B management in the interventional group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 16 years Therapeutic management within 3 hours after TBI

GCS score of 15 classically requiring hospitalization and/or CCT-scan as per SFP recommendations (Lorton et al., 2014). These criteria are:

* For children aged under 2 years (CCT-scan or hospitalization recommended according to physician's evaluation):
* Parietal or occipital scalp hematoma,
* Loss of consciousness for more than 5 seconds,
* Trauma due to serious accident (road accident with passenger ejected from vehicle or death of another person or rollover; pedestrian hit by a moving vehicle; cyclist not wearing a helmet; fall from a height greater than 0.9 meter),
* Abnormal behavior in the opinion of parents.
* For children 2 years and older (CCT-scan or hospitalization recommended according to physician's evaluation):
* Loss of consciousness at time of accident,
* Vomiting,
* Trauma due to serious accident (road accident with passenger ejected from vehicle or death of another person or rollover; pedestrian hit by a moving vehicle; cyclist not wearing a helmet; fall from a height greater than 1.5 meter),
* Severe headache.

Exclusion Criteria:

* Patient already enrolled in another therapeutic trial with drug administration Down syndrome Melanoma Refusal of child Refusal of parents or legal guardian Trauma more than 3 hours earlier GCS score of 13 or 14, or signs of skull fracture or lesions of the skull base (CCT-scan recommended)

Children with TBI not requiring hospitalization and/or CCT-scan as per SFP recommendations (Lorton et al., 2014). This group is defined by the absence of the following criteria:

* GCS score different from 15,
* Age < 3 months,
* Seriousness of accident:
* road accident with passenger ejected from vehicle or death of another person or rollover,
* pedestrian hit by a moving vehicle,
* cyclist not wearing a helmet.
* Fall:
* of more than 0.9 m before age 2 years,
* of more than 1.5 m after age 2 years.
* Loss of consciousness for 5 seconds or more,
* Inconsolable crying,
* Agitation, drowsiness, feeling "slowed down", obnubilation,
* Vomiting or headache,
* Facial or cranial hematoma,
* Otorrhea, rhinorrhea,
* Child under 2 years old,
* Loss of consciousness for less than 5 seconds,
* Unusual behaviour,
* Concern of family members

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2209 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
utility of serum S100B measurement in the management of pediatric mTBI | at day 1
  Evaluate the utility of serum S100B measurement in the management of pediatric mTBI by demonstrating a decrease in the proportion of CCT-scan prescribed in the "S100B management" intervention arm compared with the "conventional management" control arm, hypothesizing a 30% decrease in the number of CCT-scan between the intervention versus control arms.

SECONDARY OUTCOMES:
utility of serum S100B measurement with respect to reduction in the time spent in the pediatric emergency room | at day 1
utility of serum S100B measurement with respect to reduction in the duration of hospitalization | at day 1
utility of serum S100B measurement with respect to reduction in radiation exposure (mSv) | at day 1
utility of serum S100B measurement with respect to detection of complications | at day 1
  detection of complications (intracranial lesions) by CCT-scan which can occur at a rate of 0-7% in patients with mTBI (American Academy of Pediatrics, 1999)
utility of serum S100B measurement with respect to absence of intercurrent events at 48 hours and 3 weeks after mTBI | at 48 hours and 3 weeks after mTBI
utility of serum S100B measurement with respect to compliance of emergency physicians with the S100B assay | at day 1
utility of serum S100B measurement with respect to reduction of the cost of management | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Damien BOUVIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (11):
- France (11):
  - Hospices Civils de LYON, Bron
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Limoges Teaching hospital, Limoges
  - Assistance Publique des Hôpitaux de Marseille, Marseille
  - Montpellier Teaching hopsital, Montpellier
  - Nantes Teaching Hospital, Nantes
  - Nice Teaching Hospital, Nice
  - Nimes Teaching Hospital, Nîmes
  - Reims Teaching Hospital, Reims
  - Saint-Etienne Teaching Hospital, Saint-Etienne
  - Vichy Hospital Center, Vichy

REFERENCES:
- [Background] Bouvier D, Fournier M, Dauphin JB, Amat F, Ughetto S, Labbe A, Sapin V. Serum S100B determination in the management of pediatric mild traumatic brain injury. Clin Chem. 2012 Jul;58(7):1116-22. doi: 10.1373/clinchem.2011.180828. Epub 2012 Apr 23. PMID 22529109
- [Background] The management of minor closed head injury in children. Committee on Quality Improvement, American Academy of Pediatrics. Commission on Clinical Policies and Research, American Academy of Family Physicians. Pediatrics. 1999 Dec;104(6):1407-15. PMID 10585999
- [Derived] Bouvier D, Cantais A, Laspougeas A, Lorton F, Plenier Y, Cottier M, Fournier P, Tran A, Moreau E, Durif J, Sarret C, Mourgues C, Sturtz F, Oudart JB, Raffort J, Gonzalo P, Cristol JP, Masson D, Pereira B, Sapin V. Serum S100B Level in the Management of Pediatric Minor Head Trauma: A Randomized Clinical Trial. JAMA Netw Open. 2024 Mar 4;7(3):e242366. doi: 10.1001/jamanetworkopen.2024.2366. PMID 38502126
- [Derived] Bouvier D, Balayssac D, Durif J, Mourgues C, Sarret C, Pereira B, Sapin V. Assessment of the advantage of the serum S100B protein biomonitoring in the management of paediatric mild traumatic brain injury-PROS100B: protocol of a multicentre unblinded stepped wedge cluster randomised trial. BMJ Open. 2019 May 24;9(5):e027365. doi: 10.1136/bmjopen-2018-027365. PMID 31129587
- See also: Serum S100B determination in the management of pediatric mild traumatic brain injury. — http://www.ncbi.nlm.nih.gov/pubmed/22529109
- See also: The management of minor closed head injury in children. Committee on Quality Improvement, American Academy of Pediatrics. Commission on Clinical Policies and Research, American Academy of Family Physicians. — http://www.ncbi.nlm.nih.gov/pubmed/10585999